CLINICAL TRIAL: NCT06064227
Title: The Effect of Health Promotion Comprehensive Education Intervention on the Frailty Levels of Elderly Family Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fatma Banu Demirdas (Other)
Responsible Party: Sponsor-Investigator, Fatma Banu Demirdas, Principal Investigator, Akdeniz University
Organization: Akdeniz University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 3207340744
Record Dates: First submitted 2023-09-16; First posted 2023-10-03 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Frailty; Caregiver Burden; Frail Elderly Syndrome
Keywords: elderly; frailty; caregiver family members; health promotion; training intervention
MeSH Terms: conditions — Frailty; Caregiver Burden

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group. (Experimental): Multi-module training intervention.
  The intervention group, patients identified as pre-frail or frail, will be included in a multi-module educational program created specifically for this study.
  Interventions: Other: training intervention
- control group (No Intervention): The control group will be selected by single-blind, stratified randomization (coin-flip) from among patients identified as pre-frail or frail and will not receive any intervention.

INTERVENTIONS:
Other: training intervention — In this experimental study, the subject matter and sessions of the educational intervention, the effect of which was tested, were prepared based on evidence on preventable risk factors through health behavior change. The educational intervention consists of the following topics:
  Nutrition and physical exercise, chronic disease management and polypharmacy, anti-smoking and stress management, preventive health services, access to health screenings and immunization.
  Arms: intervention group.

SUMMARY:
This study was conducted to evaluate the effect of a comprehensive health promotion educational intervention applied to family caregivers over the age of 60 on their fragility levels. The main question(s) it aims to answer are:

* Does the educational intervention have a significant impact on caregivers' vulnerability?
* Does the educational intervention have a significant impact on caregivers' quality of life? The population of the study consists of family members who care for individuals receiving home health services in public hospitals in Antalya city center. G power test was used to determine the number of samples and the result of the analysis on the subject; Alpha value of 0.01 for independent sample t test at 95% confidence level; Taking an effect size of 1.35 and theoretical power of 99%, the minimum total sample size was determined as 58 people, 29 for each group. It was thought that it would be appropriate to take 30% more than the calculated minimum sample number due to possible losses that may occur during the research process, and as a result, it was decided to recruit 40 people for each group. In the study, the Participant Information Form developed by the researcher, the Health Promoting Lifestyle Profile (HPLP) scale, the frailty (FRAIL) scale and the World Health Organization quality of life scale for elderly individuals will be applied to family caregivers. SPSS statistical software package will be used in the analysis of the data obtained.

DETAILED DESCRIPTION:
While the decline in fertility rates all over the world has led to a demographic transformation, improved living conditions and technological advances have contributed to the prolongation of human life span and the increase in the number of elderly individuals. In parallel with the increase in the number of elderly people in the total population, the need for care is also increasing with long-term chronic diseases that require high-cost, complex technological intervention and care. Individuals in need of care and family caregivers prefer home care instead of institutional care for both cultural reasons and because the individual feels more autonomous at home. Therefore, the number of family members providing care at home is increasing.

Caring for family members is a stressful and time-consuming process and family caregivers are the primary caregivers of older adults. The challenges and burden of care vary depending on the circumstances and are also related to the caregiver's adaptation to the care process. The resulting maladjustment can lead to inadequate rest, interrupted sleep, chronic fatigue, economic hardship and depression, preventing the individual from meeting their own needs. Particularly if the care recipient has a cognitive impairment, the attention and time required to manage the individual's memory and behavioral issues may leave the caregiver with little time to attend to their own health needs and may neglect or delay their own care. In addition, family caregivers themselves are often elderly, chronically ill and at high risk of illness, in part due to lifestyle habits shared with the patient. All this can put caregivers at risk for emotional and physical problems and increase the susceptibility of older caregivers to health problems and frailty, a geriatric syndrome. Therefore, awareness of the risks associated with frailty, early identification and appropriate interventions can contribute to protecting and maintaining the health of this group.

The World Health Organization (WHO) has conceptually defined frailty as "a clinically recognizable condition in which older people have an increased ability to cope with daily or acute stressors due to age-related declines in physiological reserves and the functioning of multiple organ systems". Depending on the decrease in homeostatic reserves, the frailty process can be considered in three stages from non-frail to frail. These can be leveled as pre-frailty, frailty and the process of experiencing complications of frailty. Pre-frailty or fragility is clinically silent and most amenable to correction through interventions. Frailty, on the other hand, is a process in which available reserves are rapidly depleted, leading to rapid functional deterioration from well-being. The process of frailty complications can be described as an irreversible vicious circle leading to death. Although frailty has been misinterpreted in some studies as a pre-disease state that defines the end of life, the first epidemiologic data on transitions between frailty stages were reported by Gill et al (2006). Based on a 4.5-year longitudinal study of 754 older adults aged 70 years and older. In a 5-year longitudinal study of 754 older adults aged 70 years and older, it was found that 58% of participants made at least one transition between any two of the three frailty states at three follow-up visits 18 months apart, and that this transition occurred in about one-third of all visits, with participants moving from more advanced frailty states to less frailty states. This suggests that although advancing age increases the risk of frailty in individuals, frailty is not an inevitable consequence of ageing, nor is frailty an irreversible process or an inevitable path to death.

Although there is no gold standard for detecting frailty, multiple frailty screening tools have been developed and used for risk assessment and epidemiologic study. Therefore, the results of studies on the prevalence of frailty vary according to the age range, population, scale and measurement criteria used. In Europe, Eggiman et al. (2009) measured the prevalence of frailty in the same age group within the SHARE project and found the prevalence of frailty to be 17.0% and the pre-frailty rate to be 42.3%. Based on the studies in the literature, frailty risk factors can be categorized under four main headings: socio-demographic factors, lifestyle factors, medical risk factors and biological factors.

Socio-demographic factors include age, gender, ethnicity, education, low socio-economic status, living alone and loneliness, while medical risk factors include chronic diseases, multimorbidity, obesity, malnutrition, weight loss, impaired cognition, depressive symptoms and polypharmacy. Lifestyle-related risk factors include physical inactivity, diet, smoking and alcohol use. Biological risk factors include immune and neuroendocrine dysregulation, sarcopenia and energy imbalances/oxidative stress. For many individuals, the negative effects of these risk factors can be slowed down, stopped or even rapidly reversed with evidence-based early interventions for lifestyle and medical risk factors. Especially the avoidance of risky behaviors and healthy lifestyle behaviors that the individual performs with the support and awareness he/she receives have a significant contribution to the prevention of diseases and promotion of health. In the literature, there are many evidence-based studies on smoking, healthy eating, physical activity and immunization.

The onset of frailty in older people is thought to precede the behavioral adaptation that occurs in response to a reduced physiological reserve and capacity to meet environmental challenges. Xue (2011) suggested that the frailty process can be initiated through any of the clinically visible symptoms, which can then accelerate a "vicious cycle" resulting in a collective syndrome, and that different initial symptoms can lead to different rates of progression towards frailty. Recognizing and observing behavioral changes at an early stage in these older individuals, where frailty is developing but not yet detected, may be a way to intervene early in the frailty development process. Therefore, the development and evaluation of interventions designed to prevent or ameliorate frailty should be a top priority in frailty research. Pender's Health Promotion Model (HPM) is one of the most widely used models to identify and change unhealthy behaviors and improve health. This model was developed by Pender in 1987 and revised in 1996. The model guides practices in the field of health promotion and is derived from expectancy-value theory and social cognitive theory, which emphasize the importance of cognitively mediated processes in behavior choice and regulation of behavior. The Expectancy-Value Theory is based on the idea that individuals will act willingly to achieve goals whose outcomes they value, and the Social Cognitive Theory is based on the idea that individuals' thoughts direct their behaviors and that thoughts, behaviors and the environment affect each other.

The last version of the HPM, updated in 1996, consists of three main components:

1. Individual characteristics and experiences: These are biological, psychological and sociocultural factors including characteristics such as age, gender, education, income, occupation, status, personal abilities and experiences that have a direct or indirect effect on behavior.
2. Behavior-specific cognitive-perceptual factors: These are the primary motivational factors for the acquisition and maintenance of health-promoting behaviors and include perceived benefits/barriers to behaviors, perceived self-efficacy, perceived health status, mood related to the behavior, interpersonal effects and environmental-situational effects.

   Pender, assumes that perceived benefits and barriers directly affect engaging in health-promoting behaviors. Studies in the literature on the subject have revealed that older adults' participation in health promotion activities is closely related to perceived activity benefits and barriers. In terms of perceived benefits, older adults' participation in health promotion activities was found to improve their physical and psychological health, while perceived barriers were found to negatively affect their motivation in health promotion activities. The most commonly experienced barriers that prevent participation in behavior-specific health promotion activities by older adults can be defined as access barriers, lack of information, difficulty level of the health-promoting behavior, lack of social support, financial difficulties, fear of injury, and uncomfortable symptoms. Perceived Health Status, as a self-assessment of participants' perceived current overall health, is an important aspect of older adults' lives and can influence beliefs about outcomes and competencies for health-promoting behaviors. The choices an individual makes about engaging in a particular health behavior are influenced by their expectations about the outcome and beliefs about their efficacy. When an individual believes that he or she has little or no control over the outcome of a particular situation, this may prevent him or her from taking action. In Pender's Health Promotion Model, the concept of perceived self-efficacy is included as a part of cognitive and emotional factors specific to behavior. In the literature, there are many studies reporting that perceived self-efficacy is an important factor supporting an individual's participation in health promotion behaviors and lifestyle.
3. Behavior Output: This component includes making a plan for behavior; making a choice among urgent competing wants and preferences; and engaging in health behavior.

In this study, it is aimed that the educational intervention, the effect of which is to be measured, will directly or indirectly affect the "Behavior Specific Cognitive-Perceptual Factors" component defined in Pender's health model and a positive behavioral outcome will be obtained.

Gerontologists have an important position in helping caregivers accept, adapt and cope with new situations related to caregiving, while at the same time encouraging caregivers to meet their own health needs. Home caregivers need simple, practical, affordable information and advice on nutrition, chronic disease management, medication, exercise, access to health care and preventive services, and stress management. Providing these and achieving evidence-based lifestyle practices (diet and physical activity) will be an important step towards preventing frailty in this population.

ELIGIBILITY:
Inclusion Criteria:

* Being a volunteer
* Providing care to individuals with a home health service application date longer than 6 months
* Being able to speak and understand Turkish
* Being 60 years of age or older
* Having a kinship relationship with the individual they care for (mother, father, sibling, child, mother-in-law or father-in-law)

Exclusion Criteria:

* Providing care services for less than six months
* Failure to participate in one of the training modules or withdrawal from the study

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2023-09-10 (Actual)

PRIMARY OUTCOMES:
Change in total frailty score 6 months after the first educational intervention | baseline ( before intervention) and 6 months after intervention
  It consists of the sum of the scores corresponding to the participant's answers to the FRAIL scale questions.
  1. Fatigue: How much of the last 4 weeks have you felt tired? 1=Always 2=Most of the time 3=Some of the time 4=Very little of the time 5=Never (1 point if the answer is 1 or 2, 0 points for the others)
  2. Resistance: Do you have difficulty climbing 10 stairs on your own and without using an assistive device and without resting (yes: 1 point, no: 0 points)?
  3. Ambulation: "Do you have difficulty walking a few hundred meters on your own and without using an assistive device?" (1 point if yes, 0 points if no)
  4. Disease: "Has a doctor ever told you that you have the following diseases?" (Hypertension, diabetes, cancer, chronic lung disease, heart attack, congestive heart failure, angina, asthma, arthritis, stroke, kidney disease) (0-4 diseases=0 points, 5-11 diseases=1 point)
  5. Total Weight Loss within 1 year (≥5% weight loss: 1, <5% weight loss: 0)

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Banu Demirdaş, Principal Investigator
Locations (1):
- Akdeniz University, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dassel KB, Carr DC. Does Dementia Caregiving Accelerate Frailty? Findings From the Health and Retirement Study. Gerontologist. 2016 Jun;56(3):444-50. doi: 10.1093/geront/gnu078. Epub 2014 Aug 26. PMID 25161263
- [Background] Kwak D, Thompson LV. Frailty: Past, present, and future? Sports Med Health Sci. 2020 Nov 30;3(1):1-10. doi: 10.1016/j.smhs.2020.11.005. eCollection 2021 Mar. PMID 35782680
- [Background] Bhandari P, Kim M. Predictors of the Health-Promoting Behaviors of Nepalese Migrant Workers. J Nurs Res. 2016 Sep;24(3):232-9. doi: 10.1097/jnr.0000000000000120. PMID 26524721
- [Background] Hepburn M. The Variables Associated With Health Promotion Behaviors Among Urban Black Women. J Nurs Scholarsh. 2018 Jul;50(4):353-366. doi: 10.1111/jnu.12387. Epub 2018 Apr 24. PMID 29689126
- [Background] Mendis, Shanthi, et al. Global atlas on cardiovascular disease prevention and control. World Health Organization, 2011.
- [Background] Pender, N.J.; Murdaugh, C.L.; Parsons, M. Health Promotion in Nursing Practice, 6th ed.; Pearso: Boston, MA, USA, 2011; pp. 122-126.
- [Background] Gill TM, Gahbauer EA, Allore HG, Han L. Transitions between frailty states among community-living older persons. Arch Intern Med. 2006 Feb 27;166(4):418-23. doi: 10.1001/archinte.166.4.418. PMID 16505261
- [Background] Santos-Eggimann B, Cuenoud P, Spagnoli J, Junod J. Prevalence of frailty in middle-aged and older community-dwelling Europeans living in 10 countries. J Gerontol A Biol Sci Med Sci. 2009 Jun;64(6):675-81. doi: 10.1093/gerona/glp012. Epub 2009 Mar 10. PMID 19276189
- [Background] Xue QL. The frailty syndrome: definition and natural history. Clin Geriatr Med. 2011 Feb;27(1):1-15. doi: 10.1016/j.cger.2010.08.009. PMID 21093718
- [Background] Farrance C, Tsofliou F, Clark C. Adherence to community based group exercise interventions for older people: A mixed-methods systematic review. Prev Med. 2016 Jun;87:155-166. doi: 10.1016/j.ypmed.2016.02.037. Epub 2016 Feb 24. PMID 26921655